CLINICAL TRIAL: NCT00987519
Title: Viral Respiratory and Gastrointestinal Infections in Children Under 6 Years of Age - the Clinical Relevance of Newly Discovered Viruses
Brief Title: Viral Respiratory and Gastrointestinal Infections in Children Under 6 Years of Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Marko Pokorn, MD, MSc, Department of Infectious Diseases, University Medical Centre Ljubljana
Other Study IDs: VODP
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2009-10

CONDITIONS: Bronchiolitis; Gastroenteritis; Convulsion, Febrile
Keywords: acute bronchiolitis; acute gastroenteritis; febrile convulsion; viral agents; molecular methods
MeSH Terms: conditions — Bronchiolitis; Gastroenteritis; Seizures, Febrile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, stool and nasopharyngeal swab samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Acute bronchiolitis: Patients with acute bronchiolitis - the presence of nasal discharge, cough, wheezing and/or crackles on lung auscultation.
- Acute gastroenteritis: Patients with 3 or more loose or liquid stools in 24 hours prior to entering the study.
- Febrile convulsion: Patients with a cerebral paroxysm accompanied by fever without signs of central nervous system infection.
- Control group: Patients referred to pediatric surgery for elective surgical procedure - judged to be free of clinical signs and symptoms of infection.

SUMMARY:
With the use of molecular methods new viruses have been detected in respiratory and gastrointestinal tracts of both patients and asymptomatic subjects in recent years. The clinical importance of these viruses has not been adequately studied.

The aim of this study is to use molecular methods to detect viruses in upper respiratory tract and gastrointestinal tract of children with acute bronchiolitis, acute gastroenteritis and febrile convulsions and to try to correlate the severity of clinical picture with the amount of viruses present in clinical samples. The investigators will also try to detect the increase in specific antibodies in paired sera.

ELIGIBILITY:
Inclusion Criteria:

presence of

* acute bronchiolitis
* acute gastroenteritis
* febrile convulsion requiring hospital admission

Exclusion Criteria:

* none

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 6 years of age admitted to Department of Infectious Diseases, University Medical Centre Ljubljana with a diagnosis of acute bronchiolitis, acute gastroenteritis or febrile convulsion.
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To describe the clinical picture of a viral respiratory and/or gastrointestinal infection associated with a specific viral pathogen | In a 14-day period

SECONDARY OUTCOMES:
To correlate the severity of clinical picture with the quantity of virus in clinical samples | In a 14-day period

CONTACTS AND LOCATIONS:
Overall Officials: Marko Pokorn, MD, MSc, Principal Investigator — Department of Infectious Diseases, University Medical Centre Ljubljana; Franc Strle, MD, PhD, Study Chair — Department of Infectious Diseases, University Medical Centre Ljubljana; Miroslav Petrovec, MD, PhD, Principal Investigator — Institute of Microbiology and Immunology
Locations (3):
- Slovenia (3):
  - Department of Infectious Diseases, University Medical Centre Ljubljana, Ljubljana
  - Department of Pediatric Surgery, University Medical Centre Ljubljana, Ljubljana
  - Institute of Microbiology and Immunology, Ljubljana

REFERENCES:
- [Derived] Pokorn M, Jevsnik M, Petrovec M, Steyer A, Mrvic T, Grosek S, Lusa L, Strle F. Respiratory and Enteric Virus Detection in Children. J Child Neurol. 2017 Jan;32(1):84-93. doi: 10.1177/0883073816670820. Epub 2016 Oct 3. PMID 27698149
- [Derived] Jevsnik M, Steyer A, Pokorn M, Mrvic T, Grosek S, Strle F, Lusa L, Petrovec M. The Role of Human Coronaviruses in Children Hospitalized for Acute Bronchiolitis, Acute Gastroenteritis, and Febrile Seizures: A 2-Year Prospective Study. PLoS One. 2016 May 12;11(5):e0155555. doi: 10.1371/journal.pone.0155555. eCollection 2016. PMID 27171141
- [Derived] Jevsnik M, Steyer A, Zrim T, Pokorn M, Mrvic T, Grosek S, Strle F, Lusa L, Petrovec M. Detection of human coronaviruses in simultaneously collected stool samples and nasopharyngeal swabs from hospitalized children with acute gastroenteritis. Virol J. 2013 Feb 5;10:46. doi: 10.1186/1743-422X-10-46. PMID 23379823